CLINICAL TRIAL: NCT03174366
Title: Investigating the Use of Prolia (Denosumab) in the Treatment of Acute Charcot Neuroarthropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20159178
Record Dates: First submitted 2017-05-11; First posted 2017-06-02 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Charcot Joint of Foot
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Group, receiving medication (Experimental): Subjects in this group will be receiving medication (denosumab)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Subjects will receive medication once following enrollment, and will be monitored for 1 year thereafter.

SUMMARY:
Charcot neuroarthropathy (CN) is a debilitating disease primarily affecting poorly controlled diabetic patients with peripheral neuropathy. The consequences of CN include ulcerations of the foot and ankle, osteomyelitis, and severe musculoskeletal deformity. These consequences frequently lead to below-knee amputation of the affected limb.

Currently treatment options are limited, and no pharmaceutical treatment has been efficacious in the medical literature. The purpose of this pilot study is to investigate the potential of the medication denosumab for acute stage Charcot neuroarthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 30 years old
* Subject is able and willing to comply with study procedures, and is able to give signed and dated consent
* Subject meets criteria for diagnosis of Diabetes Mellitus Type 1 or 2, active Charcot neuroarthropathy, and peripheral neuropathy
* Subjects with serum calcium or albumin-adjusted serum calcium ≥2.0 mmol/L (8.0mg/dL)

Exclusion Criteria:

* Unable to provide signed and dated consent.
* Charcot neuroarthropathy of the ipsilateral lower extremity, diagnosed over 1 month prior.
* Prior foot or ankle surgery of the ipsilateral lower extremity.
* Prior amputation at any level of either lower extremity.
* Prior foot or ankle fracture of the ipsilateral lower extremity unrelated to the current acute CN episode.
* Currently has any of the following:

  1. Infection
  2. Foot ulceration
  3. Hypocalcemia
  4. Creatinine clearance less than 30 mL/min or on dialysis
  5. Pre-existing disturbance of mineral metabolism (e.g., hypoparathyroidism unstable on therapy, thyroid or parathyroid surgery, vitamin D deficiency, malabsorption syndromes, excision of small intestine, history of diseases affecting bone metabolism) that has not been effectively corrected or treated.
* Have undergone revascularization procedures of the lower extremities.
* Female subjects who are pregnant or planning to breastfeed should not participate in this study.
* Determined to have poor oral hygiene after dental screening or are at increased risk for developing osteonecrosis of the jaw.
* History of osteonecrosis of the jaw.
* History of tooth extraction or other dental surgery within the prior 6 months.
* Invasive dental work planned in the next 2 years.
* Have a known hypersensitivity to Prolia.
* Known use of a bone active medication within the 6 months prior to enrollment.
* Liver disease, defined as AST > 2.0x ULN, ALT > 2.0x ULN, TBL > 1.5x ULN.
* Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group, Receiving Medication
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 4
  Race/Ethnicity: African-American | 1
  Race/Ethnicity: Mixed Hispanic/Native American | 1
  Race/Ethnicity: Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 7
Participants
  Serious adverse event | 0
  No serious adverse events | 7

2. Secondary Outcome: Change in Skin Temperature Difference in Degrees Celsius Between the Affected and Non-affected Limb at 6 Months.
Description: Change in skin temperature difference in degrees Celsius between the affected and non-affected limb at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 7
degrees Celsius | 3.06 (0.78)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Group, Receiving Medication
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group, Receiving Medication (N=7)
Muscle pain, upper extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Injection site pain, resolved after two weeks
Cellulitis (Infections and infestations) | 1 (1) — Cellulitis of the contralateral lower extremity, resolved with oral antibiotics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT03174366/Prot_SAP_000.pdf